CLINICAL TRIAL: NCT04276298
Title: A Prospective, Multicentre, Double-Blinded Randomised Controlled Trial Comparing Topical Metronidazole, Diltiazem and Lidocaine on Post-Operative Pain Following Excisional Haemorrhoidectomy
Brief Title: Topical Analgesia Post-Haemorrhoidectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Andrew G Hill, MBChB, MD (Thesis), EdD, FACS, FRACS, Professor of Surgery, Head of School, University of Auckland, New Zealand
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RCT Haemorrhoidectomy
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Hemorrhoid Pain; Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Metronidazole; Diltiazem

STUDY DESIGN:
Intervention Model Description: Parallel with 1:1:1:1 Allocation.
Who Masked: Participant, Care Provider
Masking Description: Double blinded trial, both participant and investigator are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Metronidazole (Active Comparator): Group A receiving 10% metronidazole cream
  Interventions: Drug: Metronidazole cream
- Metronidazole + Diltiazem (Active Comparator): Metronidazole 10% + Diltiazem 2%
  Interventions: Drug: Metronidazole and Diltiazem cream
- Metronidazole + Lignocaine (Active Comparator): Metronidazole 10% + Lignocaine 4%
  Interventions: Drug: Metronidazole and Lidocaine cream
- Metronidazole + Diltiazem + Lignocaine (Active Comparator): Metronidazole 10% + Diltiazem 2% + Lignocaine 4%
  Interventions: Drug: Metronidazole, Diltiazem and Lidocaine cream

INTERVENTIONS:
Drug: Metronidazole cream — 10% metronidazole applied rectally
  Arms: Metronidazole
Drug: Metronidazole and Diltiazem cream — Combination Metronidazole and Diltiazem applied rectally
  Arms: Metronidazole + Diltiazem
Drug: Metronidazole and Lidocaine cream — Combination metronidazole and lignocaine applied rectally
  Arms: Metronidazole + Lignocaine
Drug: Metronidazole, Diltiazem and Lidocaine cream — Combination of all active agents tested applied rectally
  Arms: Metronidazole + Diltiazem + Lignocaine

SUMMARY:
Symptomatic haemorrhoids, or piles, have significant effects on quality of life. The treatment for advanced disease is surgical excision (haemorrhoidectomy) which is extremely effective. However, pain following haemorrhoidectomy is known by all to be a miserable experience and current treatment is not very effective. We have formulated a new cream treatment which targets three theorised mechanisms of pain after haemorrhoidectomy. We will test the effectiveness of the treatments with a multi-centred randomised controlled factorial trial with four parallel double-blinded arms containing different combinations of the active agents. The outcomes include pain scores, amount of analgesia required and time to return to work. The results of our study could provide evidence of an effective treatment for post haemorrhoidectomy pain. The treatment may provide considerable benefit to patients undergoing this surgical procedure.

DETAILED DESCRIPTION:
Study Design: This will be a patient-and-investigator blinded factorial randomised trial with four parallel groups. Participants in all four groups will be instructed to apply cream 3 times a day for 7 days after surgery. A standard analgesia prescription will be provided with laxatives as per routine care. Patients will be provided a questionnaire to complete and return on day 14.

Random Sequence Generation: Computer generated sequence allocating patients to a 1:1:1:1 ratio using permuted block randomisation in blocks of 12.

Allocation Concealment: This randomisation code will be seeded to the pharmacist to who will package and label the cream according to a code. The creams will be indistinguishable to which active ingredient they contain.

Assignment of intervention: Patients will be assigned in order according to the numbering of the cream tubes by the blinded investigator.

Data recording: Data will be recorded on Redcap database.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16
* All patients undergoing excisional haemorrhoidectomy

Exclusion Criteria:

* Age <16,
* history of chronic pain,
* drug allergy or idiosyncracies to any actives or excipients in
* cream,
* breastfeeding,
* any medical history which is a contraindication to any of metronidazole, lidocaine, or diltiazem including including:
* sick sinus syndrome,
* atrioventricular block,
* hypotension,
* heart failure and bradycardia.
* concomitant medications which are contraindicated to metronidazole, lidocaine or diltiazem.
* patients already taking diltiazem.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Pain scores | 7 days
  Measured by visual analog scale, 1-10cm, continuous, the higher the score, the worse the pain
Amount of analgesic use | 7 days
  Morphine equivalent amount

SECONDARY OUTCOMES:
Return to work | 14 days
  Day post-operation when the patient returns to work
Pain on bowel motion: Visual Analog Scale | 7 days
  Measured by Visual Analog Scale, continuous 1-10cm, the higher the score, the worse the pain.
Complications | 30 days
  Rates of Bleeding
Re-admission | 30 days
  Rates of Re-admission to hospital,
Repeat Prescription | 30 days
  Rates of Repeat Prescription Requirement

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hill, MBChB, MD, EdD, FRACS, FACS, Principal Investigator — Counties Manukau Health
Locations (1):
- Counties Manukau District Health Board, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Will be shared when results become available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When results are available for 12 months
Access Criteria: email request

REFERENCES:
- [Derived] Jin JZ, Xia W, Gao R, Vandal AC, Weston M, Israel L, Connolly A, Singh PP, Svirskis D, Hill A. A Randomized Controlled Trial of Topical Analgesia Posthemorrhoidectomy (TAPH Trial). Dis Colon Rectum. 2024 Sep 1;67(9):1158-1168. doi: 10.1097/DCR.0000000000003419. Epub 2024 Jun 11. PMID 38871679